CLINICAL TRIAL: NCT01258179
Title: Peri-operative Expression Analysis of Pancreatic Stone Protein and Pancreatitis-associated Protein in a Surgical Study Population
Brief Title: Peri-operative Expression Analysis of Pancreatic Stone Protein in a Surgical Study Population
Status: Terminated | Type: Observational
Why Stopped: low recruitment
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: 11.2009
Record Dates: First submitted 2010-12-07; First posted 2010-12-10 (Estimated); Last update posted 2018-05-17 (Actual); Status verified 2018-05

CONDITIONS: Patients Undergoing Major Abdominal Surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Venous blood samples
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Sepsis Group: Patients suffering from sepsis in the postoperative course after major abdominal surgery
  Interventions: Other: Analysis of PSP and PAP from venous blood samples
- Control Group: Patients without suffering sepsis during postoperative follow up after major abdominal surgery
  Interventions: Other: Analysis of PSP and PAP from venous blood samples

INTERVENTIONS:
Other: Analysis of PSP and PAP from venous blood samples — to analyse the peri-operative expression of pancreatic stone protein in surgical patients following major abdominal surgery

SUMMARY:
The purpose of this study is to analyze the peri-operative expression of pancreatic stone protein and pancreatitis-associated protein in surgical patients following major abdominal surgery by blood samples.

ELIGIBILITY:
Inclusion criteria: - >= 18 years

* abdominal major surgery
* need for post-operative ICU care

Exclusion criteria: - <18 years

- patients who do not agree the written informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing major abdominal surgery
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Diagnosed Infections according to the Systemic Inflammatory Response System (SIRS) Criteria of the german interdisciplinary Association of Intensive and Emergency Medicine | 2 years

SECONDARY OUTCOMES:
Intensive Care Unit (ICU) stay in days | 2 years
hospital stay in days | 2 years
postoperative complications according to the "Clavien-Dindo Classification" System | 2 years
hospital costs | 2 years
comparisons to other known infectious parameters: c-reactive protein (CRP), procalcitonin (PCT), Interleukin 6 (IL-6), Tumor Necrosis Factor Alpha (TNF-alpha), Leucocytes | 2 years
Bacteriaemia in the blood | 2 years
Platelets in the blood | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christian E Oberkofler, MD, Principal Investigator — UniversitaetsSpital Zuerich
Locations (1):
- Department of Visceral and Transplantation Surgery, Zurich, CH/Zürich, Switzerland

REFERENCES:
- [Derived] Fisher OM, Raptis DA, Vetter D, Novak A, Dindo D, Hahnloser D, Clavien PA, Nocito A. An outcome and cost analysis of anal fistula plug insertion vs endorectal advancement flap for complex anal fistulae. Colorectal Dis. 2015 Jul;17(7):619-26. doi: 10.1111/codi.12888. PMID 25641401
- [Derived] Fisher OM, Oberkofler CE, Raptis DA, Soll C, Bechir M, Schiesser M, Graf R. Pancreatic stone protein (PSP) and pancreatitis-associated protein (PAP): a protocol of a cohort study on the diagnostic efficacy and prognostic value of PSP and PAP as postoperative markers of septic complications in patients undergoing abdominal surgery (PSP study). BMJ Open. 2014 Mar 6;4(3):e004914. doi: 10.1136/bmjopen-2014-004914. PMID 24604486